CLINICAL TRIAL: NCT06950307
Title: Hypofractionation for Prostate Cancer in Africa: A Feasibility Study
Acronym: HypoAfrica
Status: Active, not recruiting | Type: Observational
Sponsor: Muhimbili University of Health and Allied Sciences (Other)
Collaborators: Inkosi Albert Luthuli Central Hospital (Unknown); Erasmus Medical Center (Other); Dana-Farber Cancer Institute (Other); Nigeria Sovereign Investment Authority-Lagos University Teaching Hospital Cancer Center (NLCC) (Unknown)
Responsible Party: Principal Investigator, TWALIB NGOMA, Muhimbili University College of Health Sciences Research Chair Holder, Muhimbili University of Health and Allied Sciences
Other Study IDs: HypoAfrica Prostate Cancer
Record Dates: First submitted 2025-04-15; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Radiotherapy; Hypofractionation; Africa; Acute toxicity; Late toxicity; Treatment outcome
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Low-intermediate risk: Men with localized prostate cancer - T1c-T3a, Gleason <8
  Interventions: Radiation: Hypofractionated radiotherapy for low- and intermediate-risk prostate cancer patients
- High-risk: Men with localized prostate cancer - T3b-T4 and/or Gleason ≥8
  Interventions: Radiation: Hypofractionated radiotherapy for high-risk prostate cancer patients

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy for low- and intermediate-risk prostate cancer patients — Hypofractionated radiotherapy for low- and intermediate-risk prostate cancer will be treated with 20x3 Gray (Gy), 5 days/week
  Groups: Low-intermediate risk
Radiation: Hypofractionated radiotherapy for high-risk prostate cancer patients — Hypofractionated radiotherapy for high-risk prostate cancer will be treated with 20x3.1 Gy, 5 days/week
  Groups: High-risk

SUMMARY:
Hypofractionated radiotherapy (HFRT) is a technique that delivers a higher radiation dose per treatment fraction over a shorter overall number of fractions, thus reducing the number of radiotherapy visits required to complete a course of radiation therapy. HFRT significantly alleviates the burden of transportation, accommodation, and income loss for patients while mitigating the strain on already limited healthcare personnel and infrastructure resources.

Several randomized studies conducted in Europe and the USA have demonstrated that HFRT for prostate cancer is non-inferior to conventional radiotherapy in terms of toxicity and treatment outcomes. HypoAfrica Prostate Cancer is a multi-center study that aims to explore the feasibility of implementing moderate HFRT for the treatment of localized prostate cancer in Africa. In particular, this study will evaluate the gastrointestinal and genitourinary toxicities in prostate cancer patients for up to two years post-completion of HFRT.

DETAILED DESCRIPTION:
Rationale: Radiotherapy is a critical and inseparable component of cancer treatment but access to radiotherapy is significantly inadequate in low-and middle-income countries. Adopting hypofractionated regimens as standard of care for prostate cancer offers logistical advantages by reducing the burden on the already strained radiotherapy resources in most African countries and increasing patient convenience. Several large randomized, phase 3 trials from high-income Western countries offer level I evidence to implement moderate hypofractionation for prostate cancer, providing control and toxicity similar to that of conventionally delivered fractionation. The present study will explore the feasibility of applying moderate hypofractionated radiotherapy for prostate cancer in a low- or middle- income country setting in sub-Saharan Africa.

Objective: To explore the feasibility of applying moderate hypofractionation for localized prostate cancer in an African setting.

Study design: This is a multi-centre, prospective, observational study to be conducted at 3 sites across Africa. Subject enrollment is anticipated to be completed in approximately 12 months. Subjects will be followed for up to 5 years from enrollment.

Study population: Patients with localized non-metastatic prostate cancer.

Intervention: Hypofractionated radiation therapy. Patients will be treated with 20 daily fractions, 5 times/week. Toxicity will be measured using the European Organization for Research and Treatment of Cancer-Radiation Therapy Oncology Group modified toxicity scores (EORTC-RTOG) and the Common Terminology Criteria for Adverse Events (CTCAE), version 5.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Histologically confirmed localized (low-intermediate-high risk) prostate cancer
2. Any T stage, any prostate specific antigen (PSA) value, any Gleason score, lymph node negative, non-metastatic (N0M0), based on computed tomography (CT) scan or magnetic resonance image (MRI), bone scintigraphy, and/or positron emission tomography prostate-specific membrane antigen (PET-PSMA) scan.
3. Willing to provide informed consent.
4. Willing to participate in post-treatment follow-up at 3, 12, and 24 months post-treatment.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Radiological evidence of pelvic nodal disease (CT scan, MRI, PET-PSMA scan)
2. Presence of distant metastasis (bone scintigraphy, PET-PSMA scan)
3. Patient is a candidate for elective lymph node irradiation
4. Inflammatory bowel disease
5. Previous pelvic radiotherapy
6. Previous prostatectomy
7. Bilateral hip prostheses
8. Unwilling to participate in post-treatment follow-up at 3, 12, and 24 months post-treatment

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with localized prostate cancer undergoing treatment at the trial sites
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Grade ≥2 acute gastro-intestinal and genitourinary toxicity at the end of radiotherapy | 27-30 days from start of radiotherapy
  Toxicity measured using European Organization for Research and Treatment of Cancer-Radiation Therapy Oncology Group modified toxicity scores (EORTC-RTOG) and the Common Terminology Criteria for Adverse Events (CTCAE), version 5
Cumulative grade ≥2 late gastro-intestinal and genitourinary toxicity 3-24 months after radiotherapy | 3-24 months post radiotherapy
  Toxicity measured using European Organization for Research and Treatment of Cancer-Radiation Therapy Oncology Group modified toxicity scores (EORTC-RTOG) and the Common Terminology Criteria for Adverse Events (CTCAE), version 5

SECONDARY OUTCOMES:
Any grade gastro-intestinal and genitourinary toxicity at 3-12-24 months | 3, 12, and 24 months post radiotherapy
  Toxicity measured using European Organization for Research and Treatment of Cancer-Radiation Therapy Oncology Group modified toxicity scores (EORTC-RTOG) and the Common Terminology Criteria for Adverse Events (CTCAE), version 5
PSA failure-free survival at 5 years | 5 years post-radiotherapy

OTHER OUTCOMES:
Overall survival at 5 years | 5 years post-radiotherapy
Number of patients lost-to-follow-up | 5 years post-radiotherapy

CONTACTS AND LOCATIONS:
Locations (3):
- NSIA-LUTH Cancer Center, Lagos, Lagos, Nigeria
- Inkosi Albert Luthuli Central Hospital, Durban, South Africa
- Ocean Road Cancer Institute, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Olatunji E, Swanson W, Patel S, Adeneye SO, Aina-Tofolari F, Avery S, Kisukari JD, Graef K, Huq S, Jeraj R, Joseph AO, Lehmann J, Li H, Mallum A, Mkhize T, Ngoma TA, Studen A, Wijesooriya K, Incrocci L, Ngwa W. Challenges and opportunities for implementing hypofractionated radiotherapy in Africa: lessons from the HypoAfrica clinical trial. Ecancermedicalscience. 2023 Feb 16;17:1508. doi: 10.3332/ecancer.2023.1508. eCollection 2023. PMID 37113724